CLINICAL TRIAL: NCT01195714
Title: PHASE II STUDY OF MINI-CHOP PLUS OFATUMUMAB (O) IN NON PREVIOUSLY TREATED PATIENTS AGED OVER 80 YEARS WITH CD 20+ DIFFUSE LARGE B-CELL LYMPHOMA
Brief Title: Study of Mini-Chop Plus Ofatumumab To Treat Cd 20+ Diffuse Large B-Cell Lymphoma In Patients Aged Over 80 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNH09-7B
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Non Previously Treated CD20+ Diffuse Large B-cell Lymphoma
MeSH Terms: interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab (Experimental)
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — solution for perfusion, 1000mg per cycle, 1 cycle every 3 weeks, total 6 cycles

SUMMARY:
This study is a multicentric, phase II, open-label, non-randomized trial evaluating the efficacy of O-miniCHOP in patients aged over 80 years with non previously treated CD20+ diffuse large B-cell lymphoma (age-adjusted IPI=0 to3), stage I, II, III or IV with a performance status ECOG from 0 to 4.

The anticipated study dates (start / end) are: 2010 - 2013. The study will evaluate a cohort of 120 patients (approximately 95 in France, 15 in Belgium, 5 in Switzerland and 5 in Portugal).

Patients will be recruited over 30 months and followed at least one year after the last patient has been included.

The duration of the treatment period is approximately 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patient with histologically proven CD20+ diffuse large B-cell lymphoma (DLBCL) (WHO classification 2008) including clinical subtypes (primitive mediastinal, intravascular, etc.) May also be included : de Novo Transformed DLBCL from low grade lymphoma (Follicular, other...) and DLBCL associated with some small cell infiltration in bone marrow

* Or CD20+ B-cell lymphoma, with intermediate features between DLBCL and Burkitt or with intermediate features between DLBCL and classical Hodgkin lymphoma
* Or CD20+ Follicular lymphoma grade 3B
* Or CD20+ Aggressive B-cell lymphoma unclassifiable Aged over 80 years. Ann Arbor stage I, II, III or IV. All aaIPI Patient non previously treated. All ECOG performance status With a minimum life expectancy of 3 months. Negative HIV, HBV and HCV serologies test < 4 weeks (except after vaccination). Patient able to give his consent and having previously signed a written informed consent.

Patient affiliated to social security system, if applicable

Exclusion Criteria:

Any other histological type of lymphoma, Burkitt included. Any history of treated or non-treated small-B cell lymphoma. Central nervous system or meningeal involvement by lymphoma. Contra-indication to any drug contained in the chemotherapy regimens. Any serious active disease (according to the investigator's decision). Poor renal function (creatinin level>150µmol/l), poor hepatic function (total bilirubin level>30mmol/l, transaminases>2.5 maximum normal level) unless these abnormalities are related to the lymphoma.

Poor bone marrow reserve as defined by neutrophils <1.5 G/l or platelets <100 G/l, unless related to bone marrow infiltration.

Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma. Patients previously diagnosed with prostate cancer are eligible if (1) their disease was T1-T2a, N0, M0, with a Gleason score <7, and a prostate specific antigen (PSA) <10 ng/mL prior to initial therapy, (2) they had definitive curative therapy (ie, prostatectomy or radiotherapy) >2 years before Day 1 of Cycle 1, and (3) at a minimum 2 years following therapy they had no clinical evidence of prostate cancer, and their PSA was undetectable if they underwent prostatectomy or <1 ng/mL if they did not undergo prostatectomy.

Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.

Prior treatment with anti-CD20 monoclonal antibody or alemtuzumab within 3 months prior to start of therapy Adult patient under tutelage.

Min Age: 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peyrade Frederic, MD, Study Chair — Lymphoma Study Association
Locations (84):
- Belgium (17):
  - Zna Stuivenberg, Antwerp
  - RHMS, Baudour
  - Az Sint Jan Av, Bruges
  - Institut Jules Bordet, Brussels
  - Universite Libre de Bruxelles - Hopital Erasme, Brussels
  - Ucl de Louvain St Luc, Brussels
  - Chu de Liege, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - Clinique Notre Dame de Grace, Gosselies
  - Hopital Jolimont, Haine-Saint-Paul
  - Ch Hutois, Huy
  - Az Groeninge - Campus Maria'S Voorzienigheid, Kortrijk
  - Chu Tivoli, La Louvière
  - Chr de La Citadelle, Liège
  - Clinique Saint Pierre, Ottignies
  - Universite Catholique de Louvain Mont Godinne, Yvoir
- France (67):
  - Ch Du Pays D'Aix, Aix-en-Provence
  - Ch Antibes, Antibes
  - Ch Henri Duffaut, Avignon
  - Hopital de Bayonne, Bayonne
  - Hopital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Ch Du Dr Duchenne, Boulogne-sur-Mer
  - Ch de Bour En Bresse, Bourg-en-Bresse
  - Chu de Brive, Brive-la-Gaillarde
  - Chu Cote de Nacre, Caen
  - Centre Henri Baclesse, Caen
  - Ch de Cannes, Cannes
  - Hopital de Chalon, Chalon-sur-Saône
  - Ch Chambery, Chambéry
  - Ch de Chartres - Hopital Louis Pasteur, Chartres
  - Hopital Antoine Beclere, Clamart
  - Hopital D'Instruction Des Armees Percy, Clamart
  - Hopital Pasteur, Colmar
  - Ch Compiege, Compiègne
  - Ch Sud Francilien, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - Chu Le Bocage, Dijon
  - Ch de Dunkerque, Dunkirk
  - Ch Dunkerque, Dunkirk
  - Ch Frejus St Raphael, Fréjus
  - CH GERET, Guéret
  - Hopital Saint Louis, La Rochelle
  - Hopital Andre Mignot, Le Chesnay
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - Ch de Meulan, Les Mureaux
  - Hopital St Vincent de Paul, Lille
  - Chu Claude Hurriez, Lille
  - Chu Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Chu Hopital Nord, Marseille
  - Institut Paoli Calmette, Marseille
  - Hopital Des Chanaux, Mâcon
  - Chu de Meaux, Meaux
  - Chu Marc Jacquet, Melun
  - Hopital Bon Secours, Metz
  - Crlc Val D'Aurelle - Paul Lamarque, Montpellier
  - Centre Azureen de Cancerologie, Mougins
  - Hopital Americain de Paris, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Hopital St Antoine, Paris
  - Hotel Dieu, Paris
  - Hopital St Louis, Paris
  - Hopital de La Pitie Salpetriere, Paris
  - Institut Curie, Paris
  - Hopital Necker, Paris
  - Ch Marechal Joffre, Perpignan
  - Chu Lyon Sud, Pierre-Bénite
  - Chu de Poitiers - Hopital de Miletrie, Poitiers
  - Ch Rene Dubos, Pontoise
  - Ch Annecy, Pringy
  - Chu Robert Debre, Reims
  - Ch de Roubaix - Hopital Victor Provo, Roubaix
  - Clinique Mathilde, Rouen
  - Centre Henri Becquerel, Rouen
  - Centre Rene Hugenin, Saint-Cloud
  - Ch de Saint Germain, Saint-Germain-en-Laye
  - Hopital Font Pre, Toulon
  - Chu de Toulouse, Toulouse
  - Ch de Troyes, Troyes
  - Hopital de Valence, Valence
  - Chu Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Peyrade F, Bologna S, Delwail V, Emile JF, Pascal L, Ferme C, Schiano JM, Coiffier B, Corront B, Farhat H, Fruchart C, Ghesquieres H, Macro M, Tilly H, Choufi B, Delarue R, Fitoussi O, Gabarre J, Haioun C, Jardin F. Combination of ofatumumab and reduced-dose CHOP for diffuse large B-cell lymphomas in patients aged 80 years or older: an open-label, multicentre, single-arm, phase 2 trial from the LYSA group. Lancet Haematol. 2017 Jan;4(1):e46-e55. doi: 10.1016/S2352-3026(16)30171-5. PMID 28041583